CLINICAL TRIAL: NCT02242760
Title: A Phase 2, Multi-Center, Randomized, Evaluator-Blinded, Vehicle-Controlled Study Comparing the Efficacy, Tolerability, and Safety of SB204 Gel and Vehicle Gel Once or Twice Daily in the Treatment of Acne Vulgaris
Brief Title: P2 Multi-center Study of SB204 Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-AC202
Record Dates: First submitted 2014-09-10; First posted 2014-09-17 (Estimated); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Acne Vulgaris
Keywords: acne
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- SB204 2% Twice daily (Experimental): Twice daily SB204 2%
  Interventions: Drug: SB204 2%
- SB204 4% daily (Experimental): Once daily SB204 4%
  Interventions: Drug: SB204 4%
- Vehicle Gel Daily (Placebo Comparator): Vehicle Gel Daily
  Interventions: Drug: Vehicle Gel
- Vehicle Gel Twice Daily (Placebo Comparator): Twice daily Vehicle Gel
  Interventions: Drug: Vehicle Gel
- SB204 4% Twice Daily (Experimental): Twice daily SB204 4%
  Interventions: Drug: SB204 4%

INTERVENTIONS:
Drug: SB204 2% — Applied topically twice daily
  Other Names: NVN1000
  Arms: SB204 2% Twice daily
Drug: SB204 4% — Applied topically daily
  Other Names: NVN1000
  Arms: SB204 4% Twice Daily; SB204 4% daily
Drug: Vehicle Gel — Applied topically twice and once daily
  Other Names: Placeco
  Arms: Vehicle Gel Daily; Vehicle Gel Twice Daily

SUMMARY:
This is a randomized, multi-center, double-blinded study in subjects with moderate to severe acne vulgaris. Subjects eligible to enroll will be treated once or twice daily with 2 concentrations of a topical drug in development or a vehicle. Subjects will be treated for up to 12 weeks.

DETAILED DESCRIPTION:
A randomized, multi-center, double-blinded study in subjects with moderate to severe acne vulgaris. Subjects eligible to enroll will be treated once or twice daily with 2 concentrations of a topical drug in development or a vehicle. Subjects will be treated for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe acne
* 25-70 non-inflammatory lesions at Baseline
* 20-40 inflammatory lesions at Baseline

Exclusion Criteria:

* Subjects with known allergy to any component of the test material or vehicle
* Women who are pregnant or nursing

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 213 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M J Rico, MD, Study Director — Novan, Inc.
Locations (20):
- United States (20):
  - Qst acne site #1, Hot Springs, Arkansas
  - QST Site #118, Encinitas, California
  - QST Site #111, San Diego, California
  - QST Site #113, San Diego, California
  - QST Site #119, Santa Monica, California
  - QST Site #103, Boca Raton, Florida
  - QST Site # 110, Pinellas Park, Florida
  - QST Site # 116, Newnan, Georgia
  - QST Site #117, Louisville, Kentucky
  - QST Site #112, Detroit, Michigan
  - QST Site #120, Warren, Michigan
  - QST Site # 121, Minneapolis, Minnesota
  - QST Site #107, New York, New York
  - QST Site #108, Rochester, New York
  - QST Site #109, Rochester, New York
  - QST Site #104, Stony Brook, New York
  - QST Site # 102, San Antonio, Texas
  - QST Site #106, Salt Lake City, Utah
  - QST #105, Lynchburg, Virginia
  - QST Site #114, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle Gel QD: Vehicle Gel: Applied topically once daily
- Vehicle Gel BID: Vehicle Gel: Applied topically twice daily
- SB204 2% BID: SB204 2%: Applied topically twice daily
- SB204 4% QD: SB204 4%: Applied topically once daily
- SB204 4% BID: SB204 4%: Applied topically twice daily
Period: Overall Study
Arm/Group | Vehicle Gel QD | Vehicle Gel BID | SB204 2% BID | SB204 4% QD | SB204 4% BID
Started | 27 | 29 | 53 | 52 | 52
Number of Subjects Excluded From ITT Population (One subject in the SB204 4% BID group was not dispensed study medication after randomization.) | 0 | 0 | 0 | 0 | 1
Completed | 24 | 20 | 51 | 48 | 48
Not Completed | 3 | 9 | 2 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population: all study subjects who were randomized and dispensed study medication. One subject in the SB204 4% BID group was randomized but did not receive study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Gel QD | Vehicle Gel BID | SB204 2% BID | SB204 4% QD | SB204 4% BID | Total
Number analyzed (Participants) | 27 | 29 | 53 | 52 | 51 | 212
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Statistical Analysis Plan specified that demographic data would be presented by the individual cohorts, the combined SB204 cohorts and the combined vehicle cohort. For the SB204 cohorts, columns 3, 4, and 5 represent the individual cohorts, while column 6 represents the combined SB204 information. The individual vehicle gel cohorts are presented in columns 1 and 2, while the combined vehicle gel cohort information is in column 6.
  years
    SB204: number analyzed (Participants) | 0 | 0 | 53 | 52 | 51 | 156
    SB204 |  |  | 20.1 (6.81) | 18.8 (5.00) | 20.1 (6.94) | 19.6 (6.30)
    Vehicle: number analyzed (Participants) | 27 | 29 | 0 | 0 | 0 | 56
    Vehicle | 16.7 (4.84) | 19.7 (6.33) |  |  |  | 18.2 (5.81)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Statistical Analysis Plan specified that demographic data would be presented by the individual cohorts, the combined SB204 cohorts and the combined vehicle cohort. For the SB204 cohorts, columns 3, 4, and 5 represent the individual cohorts, while column 6 represents the combined SB204 information. The individual vehicle gel cohorts are presented in columns 1 and 2, while the combined vehicle gel cohort information is in column 6.
  Participants
    SB204: number analyzed (Participants) | 0 | 0 | 53 | 52 | 51 | 156
    SB204: Female |  |  | 26 | 29 | 29 | 84
    SB204: Male |  |  | 27 | 23 | 22 | 72
    Vehicle: number analyzed (Participants) | 27 | 29 | 0 | 0 | 0 | 56
    Vehicle: Female | 11 | 16 |  |  |  | 27
    Vehicle: Male | 16 | 13 |  |  |  | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Statistical Analysis Plan specified that demographic data would be presented by the individual cohorts, the combined SB204 cohorts and the combined vehicle cohort. For the SB204 cohorts, columns 3, 4, and 5 represent the individual cohorts, while column 6 represents the combined SB204 information. The individual vehicle gel cohorts are presented in columns 1 and 2, while the combined vehicle gel cohort information is in column 6.
  Participants
    SB204: number analyzed (Participants) | 0 | 0 | 53 | 52 | 51 | 156
    SB204: Hispanic or Latino |  |  | 13 | 10 | 9 | 32
    SB204: Not Hispanic or Latino |  |  | 40 | 42 | 42 | 124
    SB204: Unknown or Not Reported |  |  | 0 | 0 | 0 | 0
    Vehicle: number analyzed (Participants) | 27 | 29 | 0 | 0 | 0 | 56
    Vehicle: Hispanic or Latino | 4 | 4 |  |  |  | 8
    Vehicle: Not Hispanic or Latino | 23 | 25 |  |  |  | 48
    Vehicle: Unknown or Not Reported | 0 | 0 |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Statistical Analysis Plan specified that demographic data would be presented by the individual cohorts, the combined SB204 cohorts and the combined vehicle cohort. For the SB204 cohorts, columns 3, 4, and 5 represent the individual cohorts, while column 6 represents the combined SB204 information. The individual vehicle gel cohorts are presented in columns 1 and 2, while the combined vehicle gel cohort information is in column 6.
  Participants
    SB204: number analyzed (Participants) | 0 | 0 | 53 | 52 | 51 | 156
    SB204: American Indian or Alaska Native |  |  | 0 | 0 | 0 | 0
    SB204: Asian |  |  | 2 | 3 | 3 | 8
    SB204: Native Hawaiian or Other Pacific Islander |  |  | 1 | 2 | 0 | 3
    SB204: Black or African American |  |  | 9 | 6 | 10 | 25
    SB204: White |  |  | 41 | 36 | 36 | 113
    SB204: More than one race |  |  | 0 | 5 | 2 | 7
    SB204: Unknown or Not Reported |  |  | 0 | 0 | 0 | 0
    Vehicle: number analyzed (Participants) | 27 | 29 | 0 | 0 | 0 | 56
    Vehicle: American Indian or Alaska Native | 0 | 0 |  |  |  | 0
    Vehicle: Asian | 0 | 0 |  |  |  | 0
    Vehicle: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  | 0
    Vehicle: Black or African American | 4 | 5 |  |  |  | 9
    Vehicle: White | 23 | 21 |  |  |  | 44
    Vehicle: More than one race | 0 | 3 |  |  |  | 3
    Vehicle: Unknown or Not Reported | 0 | 0 |  |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: The SAP specified that demographic data would be presented by the individual cohorts, the combined SB204 cohorts and the combined vehicle cohort. The SB204 cohorts are presented in Row 1--columns 3, 4, and 5 represent the individual SB204 cohorts, while column 6 represents the combined SB204 cohort. The vehicle gel cohorts are presented in Row 2. The individual vehicle cohorts are presented in columns 1 and 2, while the combined vehicle gel cohort information is in column 6.
  Participants
    United States: SB204 | 0 | 0 | 53 | 52 | 51 | 156
    United States: Vehicle | 27 | 29 | 0 | 0 | 0 | 56

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Inflammatory Lesion Counts
Description: Change in inflammatory lesion count from Baseline to Week 12
Time Frame: Baseline and Week 12
Population: Intent to treat population (ITT)
Measure: Mean (Standard Deviation); unit: inflammatory acne lesions
Arm/Group | Vehicle Gel QD | Vehicle Gel BID | SB204 2% BID | SB204 4% QD | SB204 4% BID
Number analyzed (Participants) | 27 | 29 | 53 | 52 | 51
inflammatory acne lesions | -7.7 (10.51) | -4.1 (12.77) | -11.2 (9.48) | -11.3 (9.66) | -10.4 (9.65)

2. Primary Outcome: Absolute Change in Non-inflammatory Lesion Counts
Description: Absolute Change in non-inflammatory lesion count from Baseline to Week 12
Time Frame: Baseline and Week 12
Population: Intent to treat (ITT) population
Measure: Mean (Standard Deviation); unit: non-inflammatory acne lesions
Arm/Group | Vehicle Gel QD | Vehicle Gel BID | SB204 2% BID | SB204 4% QD | SB204 4% BID
Number analyzed (Participants) | 27 | 29 | 53 | 52 | 51
non-inflammatory acne lesions | -8.4 (16.16) | -6.9 (18.16) | -12.3 (14.91) | -14.1 (15.13) | -11.1 (17.65)

3. Primary Outcome: Proportion of Success According to the Dichotomized Investigator Global Assessment [IGA] at End of Treatment
Description: Proportion of subjects at end of treatment achieving IGA of 'clear' or 'almost clear' and a change of at least 2 in the IGA from baseline. The IGA was a static assessment. The assessment was made with the evaluator approximately 3 feet away from the subject; the IGA assessment was to be done prior to the lesion counts. A lower grade is considered to be a better outcome.
  Grade 0 = clear (clear skin with no inflammatory or non-inflammatory lesions) Grade 1 = almost clear (few non-inflammatory lesions with no more than rare papules (papules may be resolving and hyperpigmented, though not pink-red) Grade 2 = mild (some non-inflammatory lesions with no more than a few inflammatory lesions) Grade 3 = moderate (up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than 1 nodular lesion) Grade 4= severe (up to many non-inflammatory and inflammatory lesions, including nodular lesions)
Time Frame: Baseline and Week 12
Population: Intent to treat (ITT) population. Count of participants = number of participants achieving success on the Investigator's Global Assessment at Week 12: a score of clear (0) or almost clear (1) and at least 2 grades less than Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Gel QD | Vehicle Gel BID | SB204 2% BID | SB204 4% QD | SB204 4% BID
Number analyzed (Participants) | 27 | 29 | 53 | 52 | 51
Participants | 2 | 2 | 8 | 6 | 7

4. Secondary Outcome: Percent Change in Inflammatory Lesion Count From Baseline to Week 12
Description: The percent change in inflammatory lesion count from Baseline to Week 12
Time Frame: Baseline and Week 12
Population: Intent to treat (ITT) population
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Vehicle Gel QD | Vehicle Gel BID | SB204 2% BID | SB204 4% QD | SB204 4% BID
Number analyzed (Participants) | 27 | 29 | 53 | 52 | 51
Percentage change from baseline | -26.2 (34.78) | -12.5 (48.25) | -41.9 (31.35) | -41.6 (36.6) | -42.1 (35.12)

5. Secondary Outcome: Percent Change in Non-inflammatory Lesion Count From Baseline to Week 12
Description: The percent change in non-inflammatory lesion count from Baseline to Week 12
Time Frame: Baseline and Week 12
Population: Intent to treat (ITT) population
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Vehicle Gel QD | Vehicle Gel BID | SB204 2% BID | SB204 4% QD | SB204 4% BID
Number analyzed (Participants) | 27 | 29 | 53 | 52 | 51
Percentage change from baseline | -20.2 (42.54) | -14.3 (54.10) | -33.8 (33.91) | -36.8 (35.54) | -33.0 (40.16)

6. Secondary Outcome: Median Time to Improvement
Description: Median time to a 35% improvement in inflammatory lesion counts (Kaplan-Meier estimate). The full range values presented below are estimates made from the Kaplan-Meier figure.
Time Frame: Baseline through Week 12
Population: Intent to treat (ITT) population. The vehicle QD and vehicle BID arms were combined per the study Statistical Analysis Plan: "Median time to improvement will be calculated using the Kaplan-Meier method, and the Kaplan-Meier curves will be presented for each active treatment group and the combined Vehicle group."
Measure: Median (Full Range); unit: Weeks
Groups:
- Combined Vehicle: Vehicle Gel applied once or twice daily according to randomization
Arm/Group | Combined Vehicle | SB204 2% BID | SB204 4% QD | SB204 4% BID
Number analyzed (Participants) | 56 | 53 | 52 | 51
Weeks | 11.6 [1.4 to 12.1] | 2.0 [2.0 to 14] | 4.1 [1.7 to 12.3] | 4.0 [1.6 to 12]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time the subject signed the Informed Consent Form until the final study visit; an average of 12 weeks. Treatment emergent adverse events were those with an onset on or after the date of the first application of study medication. Adverse events noted prior to the first study drug administration that worsened after Baseline were also reported as AEs.
Arm/Group | Vehicle Gel QD | Vehicle Gel BID | SB204 2% BID | SB204 4% QD | SB204 4% BID
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/29 | 0/53 | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/29 | 0/53 | 1/52 | 0/51
Other Adverse Events (participants affected / at risk) | 1/26 | 4/29 | 4/53 | 5/52 | 3/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Gel QD (N=26) | Vehicle Gel BID (N=29) | SB204 2% BID (N=53) | SB204 4% QD (N=52) | SB204 4% BID (N=51)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Event required hospitalization; considered unlikely to be related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Gel QD (N=26) | Vehicle Gel BID (N=29) | SB204 2% BID (N=53) | SB204 4% QD (N=52) | SB204 4% BID (N=51)
Application site dryness (General disorders) | 0 | 0 | 0 | 3 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 3 | 2 | 1
Headache (Nervous system disorders) | 0 | 2 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2014-10-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT02242760/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT02242760/SAP_001.pdf